CLINICAL TRIAL: NCT02047669
Title: Implementation of Physical Exercise at the Workplace (IRMA09) - Laboratory Technicians
Acronym: IRMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Collaborators: University of Southern Denmark (Other); University of Southampton (Other)
Responsible Party: Principal Investigator, Lars L. Andersen, Professor, PhD, National Research Centre for the Working Environment, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRMA09
Record Dates: First submitted 2014-01-26; First posted 2014-01-28 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Musculoskeletal Disorders; Stress
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Models, Biopsychosocial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biopsychosocial (Experimental): Biopsychosocial intervention with Individually tailored physical exercises and stress management
  Interventions: Behavioral: Biopsychosocial
- Reference (Active Comparator): Reference group receiving "usual care" in terms of standard workplace ergonomics and physical exercises
  Interventions: Behavioral: Reference

INTERVENTIONS:
Behavioral: Biopsychosocial
  Arms: Biopsychosocial
Behavioral: Reference
  Arms: Reference

SUMMARY:
Musculoskeletal disorders and stress of employees remain a major problem in many occupations. The aim of this study is to investigate the effect of an individually tailored bio-psycho-social intervention strategy versus "usual care" ergonomics and standard physical exercises (reference group) on musculoskeletal pain, work disability, and stress in lab technicians with a history of work-related musculoskeletal pain.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory technician
* Pain intensity >= 3 (scale of 0-10)
* Pain duration >= 3 months
* Pain frequency >= 3 days per week

Exclusion Criteria:

* life threatening disease
* pregnancy

Ages: 18 Years to 67 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pain intensity | change from baseline to week 10
  The change in "pain intensity during the last week" (average value of back, neck, shoulder, elbow and hand) from baseline to 10 week follow-up between the individually tailored biopsychosocial group and reference group. 2-way analysis of variance with repeated measures will be used, with time, group and time x group as fixed factors and subject as random factor. Analyses will be controlled for pain intensity at baseline.

SECONDARY OUTCOMES:
Stress | change from baseline to week 10
  Cohens perceived stress scale

OTHER OUTCOMES:
WAI | change from baseline to week 10
  Work ability index questionnaire
Fear Avoidance | change from baseline to week 10
  Fear avoidance is evaluated by the Fear Avoidance Beliefs questionnaire (FABQ) by Waddell et al. at baseline and follow-up. Briefly, the FABQ is a two-part questionnaire. The first part consists of five questions/statements about pain and physical activity and the second part consists of 11 questions/statements about how work affects the participants' perception of pain. Each question is scored from 0-5 ranging from completely disagree (0) to completely agree (5).
Muscle function | change from baseline to week 10
  Muscle strength, function and tenderness of the shoulder, arm, wrist/hand is assessed by maximal isometric voluntary contractions in a custom-built dynamometer (Bofors Elektronik, Karlskoga, Sweden) setting and by pressure-pain threshold testing (PPT). Also rate of force development (RFD), force steadiness (FS), force precision (FP) and fatigue (F) are measured by using custom-made MATLAB programs. The strength tests are a part of an extensive physical examination by trained (and blinded) medical professionals at baseline and follow-up. Muscle activation level is measured by surface electromyography (EMG) (Nexus Mark 10, Mindmedia, Netherlands) on the forearm extensors, shoulder external rotator (Infraspinatus Mm.) and descending part of the trapezius muscle. Further, surface EEG (Nexus Mark 10, Mindmedia, Netherlands) will measure global brain activity during pre- and post testing by using a single a single sensor placement on the forehead (Fpz).

CONTACTS AND LOCATIONS:
Overall Officials: Lars L Andersen, PhD, Principal Investigator — National Research Centre for the Working Environment, Denmark
Locations (1):
- National Research Centre for the Working Environment, Copenhagen, Denmark

REFERENCES:
- [Derived] Jay K, Brandt M, Hansen K, Sundstrup E, Jakobsen MD, Schraefel MC, Sjogaard G, Andersen LL. Effect of Individually Tailored Biopsychosocial Workplace Interventions on Chronic Musculoskeletal Pain and Stress Among Laboratory Technicians: Randomized Controlled Trial. Pain Physician. 2015 Sep-Oct;18(5):459-71. PMID 26431123
- [Derived] Jay K, Brandt M, Sundstrup E, Schraefel M, Jakobsen MD, Sjogaard G, Andersen LL. Effect of individually tailored biopsychosocial workplace interventions on chronic musculoskeletal pain, stress and work ability among laboratory technicians: randomized controlled trial protocol. BMC Musculoskelet Disord. 2014 Dec 18;15:444. doi: 10.1186/1471-2474-15-444. PMID 25519844